CLINICAL TRIAL: NCT00893516
Title: A Multicentre Open-label Dose Escalation Tiral of Zanolimumab in Combination With CHOP Chemotherapy in Patients With CD4 Positive Non-cutaneous Peripheral T-cell Lymphoma With Nodal Involvement.
Brief Title: CD4 in Combination With CHOP in Treating Non-cutaneous Peripheral TCell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Portfolio consolidation.
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN112
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: T-cell Lymphoma
Keywords: non cutaneous peripheral t-cell lymphoma with nodal involvement
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CHOP chemo therapy + CD4 therapy
  Interventions: Biological: CHOP + CD4
- 2 (Active Comparator): CHOP chemotherapy
  Interventions: Drug: CHOP

INTERVENTIONS:
Biological: CHOP + CD4
  Arms: 1
Drug: CHOP
  Arms: 2

SUMMARY:
Evaluation of CD4 in combination with CHO chemotherapy in subjects with nodal involvement of non cutaneous Tcell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* study is closed to enrollment

Exclusion Criteria:

* study is closed to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All efforts to obtain data have been exhausted, therefore we have no data available to report.
Groups:
- 1 CHOP Chemo Therapy + CD4 Therapy CHOP + CD4: CHOP chemo therapy + CD4 therapy
  CHOP + CD4
- 2 CHOP Chemotherapy CHOP: CHOP chemotherapy
  CHOP
Period: Overall Study
Arm/Group | 1 CHOP Chemo Therapy + CD4 Therapy CHOP + CD4 | 2 CHOP Chemotherapy CHOP
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All efforts to obtain data have been exhausted, therefore we have no data available to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 CHOP Chemo Therapy + CD4 Therapy CHOP + CD4 | 2 CHOP Chemotherapy CHOP | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Unavailable
Description: All efforts to obtain data have been exhausted, therefore we have no data available to report.
Population: All efforts to obtain data have been exhausted, therefore we have no data available to report.
Arm/Group | 1 CHOP Chemo Therapy + CD4 Therapy CHOP + CD4 | 2 CHOP Chemotherapy CHOP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All efforts to obtain data have been exhausted, therefore we have no data available to report.
Arm/Group | 1 CHOP Chemo Therapy + CD4 Therapy CHOP + CD4 | 2 CHOP Chemotherapy CHOP
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
All efforts to obtain data have been exhausted, therefore we have no data available to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No